CLINICAL TRIAL: NCT06903754
Title: Sodium Glucose Cotransporter 2 Inhibitors in Patients Without Diabetes With Acute Coronary Syndrome Undergoing Percutaneous Coronary Intervention
Brief Title: ISGLT2 in Patients Without DM With Acute MI
Acronym: ISGTL2-MORMI
Status: Completed | Type: Observational
Sponsor: Mohammed VI University Hospital (Other)
Responsible Party: Principal Investigator, BOUCHLARHEM AMINE, CLINICAL CARDIOLOGIST, Mohammed VI University Hospital
Other Study IDs: DI657483
Record Dates: First submitted 2025-03-22; First posted 2025-04-01 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Acute Coronary Syndromes; Heart Failure
Keywords: Acute coronary syndronme; ISGLT2; Heart failure
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Without ISGLT2: Patients for whom we will not prescribe ISGLT2
  Interventions: Drug: With ISGLT2

INTERVENTIONS:
Drug: With ISGLT2 — Patients for whom we will prescribe ISGLT2

SUMMARY:
This study will evaluate the effect of ISGLT2 (Dapagliflozin or Empalgliflozin), administered once daily in addition to standard of care treatments for non-diabetic patients with myocardial infarction (MI) treated with PCI, on hospitalization for heart failure, readmissions for acute coronary syndrome and all-cause mortality.

DETAILED DESCRIPTION:
This is a single-center, prospective study in non-diabetic patients with acute coronary syndrome (ACS) (ST elevation (STEMI) or non-ST elevation (NSTEMI) with left ventricular systolic dysfunction (Defined as Ejection Fraction<50% assessed by 2D Simson Bi-plane echocardiography) or evidence of acute de Novo heart failure. The study will assess the effect of dapagliflozin or empagliflozin versus placebo, administered once daily in addition to standard therapy, on HF hospitalizations, all-cause deaths and ACS readmissions.

ELIGIBILITY:
Inclusion Criteria :

* Participant must approved the informed consent.
* Confirmed MI, either STEMI or NSTEMI, according to the fourth universal definition of MI (Thygesen et al 2019).
* Evidence of impaired regional or global LV systolic function at any timepoint during current MI-related hospitalisation with Ejection Fraction<50%(established with echocardiogram, radionuclide ventriculogram, contrast angiography or cardiac MRI) or Symptoms of Acute heart failure without cardiogenic Shock.
* Hemodynamically stable (no episodes of symptomatic hypotension, or arrhythmia with haemodynamic compromise in the last 24 hours).

Exclusion Criteria:

* Known type 1 diabetes mellitus (T1DM) or T2DM at the time for admission.
* Chronic symptomatic HF with a prior HHF within the last year and known reduced ejection fraction (LVEF≤40 %), documented before the current MI hospitalization.
* Patients with cardiogenic shock who received vasoactive drugs during index.
* Hospitalization Severe (eGFR <20 mL/min/1.73 m2 by local laboratory), unstable or rapidly progressing renal disease at the time of randomization
* Severe hepatic impairment (Child-Pugh class C) at the time of inclusion into the trial.
* Active malignancy requiring treatment at the time of screening.
* Any non-CV condition, eg malignancy, with a life expectancy of less than one years based on the investigator´s clinical judgement.
* Currently on treatment, or with an indication for treatment, with a sodium glucose co-transporter 2 inhibitor (SGLT2-inhibitor)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with Acute coronary syndrome
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Primary endpoints | 50 months
  Time to the first occurrence of any of the components of this composite: hospitalization for heart failure (HHF), Non fatal Myocardial infarction (MI) or Death from all causes

SECONDARY OUTCOMES:
Secondary outcomes | 50 months
  Time to the first occurrence of a fatal or a non-fatal MI [Time Frame: From admission visit (Day 0) up to approximately 4.2years] Time to first hospitalisation for Heat failure [Time Frame: From admission visit (Day 0) up to approximately 3 years] Time to death of any cause [Time Frame: From admission visit (Day 0) up to approximately 4.2 years] Time to new onset of type 2 diabetes mellitus (T2DM) post discharge [Time Frame: From admission (Day 0) up to approximately 4.2 years] Time to new onset atrial fibrilation (AF) post discharge [Time Frame: From admission visit (Day 0) up to approximately 4.2 years]

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed VI university hospital oujda, OUDA, Morocco

IPD SHARING:
Plan to Share IPD: Undecided